CLINICAL TRIAL: NCT05290636
Title: Communication Competence and Transdisciplinary Cooperation in Geriatric Nursing: A Participatory Action Research
Brief Title: Communication Competence and Transdisciplinary Cooperation in Geriatric Nursing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Chia Jung Hsieh, Ph.D., RN, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FJU-IRB C107105
Record Dates: First submitted 2022-03-03; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Communication; Competence
Keywords: Geriatric Nursing; Communication; Cooperation; Competency; Action Research
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm trial (Experimental): A single-arm trial was designed. (Two-hour sessions per week for 18 weeks). The value of classroom learning and practical experience for the study subjects is emphasized in this intervention course. The case analysis teaching technique will be used extensively in the classroom, and the school's digital action learning platform will support instructional activities relevant to senior nursing and elderly nursing practice. In each section of the course, combine classroom instruction with case analysis (2 hours each, 20-30 minutes for topic teaching, 70-80 minutes for case discussion and feedback)
  Interventions: Other: Teaching intervention program

INTERVENTIONS:
Other: Teaching intervention program — Using an action research approach, The investigators designed a pair of geriatric nursing and practicum courses and recruited a class of in-service nursing students through convenience sampling in a college setting. The intervention was an 18-week course in geriatric nursing that meets once a week in the classroom and internship practice in settings used for training nursing students. The investigators collected data using quantitative indicators (attitude measurements) and qualitative textual analysis. The quantitative data were analyzed by paired t-testing using SPSS 21.0 software.

SUMMARY:
The ability to communicate and cooperate effectively is essential in geriatric nursing. However, nursing teachers lacked the exploration of the development of this ability and teaching evaluation in previous studies. The investigators used a systematic process to investigate methods for achieving the following goals: 1. Cultivate a positive attitude toward the elderly among nursing students. 2. Improve nursing students' communication competence and interaction skills when providing advanced health care services. 3. Improve the teaching skills of professional nursing instructors.

DETAILED DESCRIPTION:
The ability to communicate and cooperate effectively is essential in geriatric nursing. However, nursing teachers lacked the exploration of the development of this ability and teaching evaluation in previous studies. The investigators used a systematic process to investigate methods for achieving the following goals: 1. Cultivate a positive attitude toward the elderly among nursing students. 2. Improve nursing students' communication competence and interaction skills when providing advanced health care services. 3. Improve the teaching skills of professional nursing instructors.

Using an action research approach, the investigators designed a pair of geriatric nursing and practicum courses and recruited a class of in-service nursing students through convenience sampling in a college setting. The intervention was an 18-week course in geriatric nursing that meets once a week in the classroom and internship practice in settings used for training nursing students. The investigators collected using quantitative indicators (attitude measurements) and qualitative textual analysis. The quantitative data were analyzed by paired t-testing using SPSS 21.0 software.

ELIGIBILITY:
Inclusion Criteria:

* The research object of this project will be the students in the nursing class of a university (third year students), and the students who have taken 2 credits each of "Geriatric Nursing" and "Geriatric Nursing Internship" in a working class.

Exclusion Criteria:

* Not a junior in a working class in a university nursing department.Those who have not completed the courses of "Geriatric Nursing" and "Geriatric Nursing Internship".

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Scale of attitudes towards the elderly | Baseline (T0)
  The scale of attitude towards the elderly is divided into positive and negative attitudes, with 20 and 22 questions respectively. This scale uses a visual analogue scale (VAS) from 1 to 7 points, ranging from From 1="strongly disagree" to 7="strongly agree", check the attitude and feeling that most matches with them. Degree detection (Cronach's α=0.94) has good reliability and validity.
Attitude Inventory for Health Team Care | Baseline (T0)
  The attitude scale of health team care, the subjects will choose the most consistent attitude and feeling from 1="strongly disagree" to 6="strongly agree" with regard to the degree of agreement between the declarative sentences and their own feelings. The higher the score of the total scale, the more positive the attitude towards health care, and the content validity of this scale has been reviewed by experts. The degree of detection (Cronach's α=0.78), so this research tool also has good reliability and validity.
Scale of attitudes towards the elderly | Change from after intervention at eighteen weeks (T1)
  The scale of attitude towards the elderly is divided into positive and negative attitudes, with 20 and 22 questions respectively. This scale uses a visual analogue scale (VAS) from 1 to 7 points, ranging from From 1="strongly disagree" to 7="strongly agree", check the attitude and feeling that most matches with them. Degree detection (Cronach's α=0.94) has good reliability and validity.
Attitude Inventory for Health Team Care | Change from after intervention at eighteen weeks (T1)
  The attitude scale of health team care, the subjects will choose the most consistent attitude and feeling from 1="strongly disagree" to 6="strongly agree" with regard to the degree of agreement between the declarative sentences and their own feelings. The higher the score of the total scale, the more positive the attitude towards health care, and the content validity of this scale has been reviewed by experts. The degree of detection (Cronach's α=0.78), so this research tool also has good reliability and validity.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Jung Hsieh, PhD, Principal Investigator — 365,Ming-te Road,Peitou District,Taipei City
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barba BE, Gendler P. Education/community collaborations for undergraduate nursing gerontological clinical experiences. J Prof Nurs. 2006 Mar-Apr;22(2):107-11. doi: 10.1016/j.profnurs.2006.01.008. PMID 16564476
- [Result] de Almeida Tavares JP, da Silva AL, Sa-Couto P, Boltz M, Capezuti E. Portuguese nurses' knowledge of and attitudes toward hospitalized older adults. Scand J Caring Sci. 2015 Mar;29(1):51-61. doi: 10.1111/scs.12124. Epub 2014 Mar 13. PMID 24628017
- [Result] Hsieh PL, Chen CM. Nursing Competence in Geriatric/Long Term Care Curriculum Development for Baccalaureate Nursing Programs: A Systematic Review. J Prof Nurs. 2018 Sep-Oct;34(5):400-411. doi: 10.1016/j.profnurs.2018.05.006. Epub 2018 Jun 1. PMID 30243697
- [Result] Ironside PM, Tagliareni ME, McLaughlin B, King E, Mengel A. Fostering geriatrics in associate degree nursing education: an assessment of current curricula and clinical experiences. J Nurs Educ. 2010 May;49(5):246-52. doi: 10.3928/01484834-20100217-01. PMID 20210290
- [Result] Mezey M, Boltz M, Esterson J, Mitty E. Evolving models of Geriatric Nursing care. Geriatr Nurs. 2005 Jan-Feb;26(1):11-5. doi: 10.1016/j.gerinurse.2004.11.012. PMID 15716809
- [Result] Rosenfeld P, Bottrell M, Fulmer T, Mezey M. Gerontological nursing content in baccalaureate nursing programs: findings from a national survey. J Prof Nurs. 1999 Mar-Apr;15(2):84-94. doi: 10.1016/s8755-7223(99)80079-9. PMID 10194893
- [Result] Yanamadala M, Kaprielian VS, O'Connor Grochowski C, Reed T, Heflin MT. A problem-based learning curriculum in geriatrics for medical students. Gerontol Geriatr Educ. 2018 Apr-Jun;39(2):122-131. doi: 10.1080/02701960.2016.1152268. Epub 2016 Sep 16. PMID 26909895